CLINICAL TRIAL: NCT06716619
Title: A Phase I Clinical Trial of the Safety and Tolerability of Tumor-Associated Lymph Node T-Cell Injection (TAL-T) in Subjects With Advanced Malignant Solid Tumors
Brief Title: A Phase I Trial of Tumor-Associated Lymph Node T-Cell Injection With Advanced Malignant Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Guangzhou FineImmune Biotechnology Co., LTD. (Industry)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIT003-001
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Tumor Associated Lymph Node T Cell; Advanced Solid Tumor; Immunotherapy; Serplulimab Injection
Keywords: Immunotherapy; Advanced Solid Tumor; Tumor Associated Lymph Node T Cell; TAL-T; cell therapy; Serplulimab Injection; Adverse Drug Event; Efficacy; Safety
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exploration of the dosage range and Expansion phase (Experimental): In the exploration dosage range phase, the safety data accumulated from the trial will be used to evaluate whether the safety of TAL-T cell therapy meets the requirements and decide whether to terminate the study. Exploration of the dosage range is divided into three dose phases, and the upper limit of the maximum dose is constantly expanded.
  After completion of exploration study, three types of preferred tumor will be choosed by sponsor. During the expansion phase, the actual number of participants in each cohort may be adjusted based on the obtained trial results to further evaluate the safety, tolerability, and efficacy of TAL-T cell infusion.
  Interventions: Biological: Tumor Associated Lymph node T cell; Drug: Serplulimab Injection

INTERVENTIONS:
Biological: Tumor Associated Lymph node T cell — At least one lymph sample is resected from each participant, then it is separated and cultured ex vivo to expand the population of Tumor Associated Lymph node T cells . After lymphodepletion, patients are infused with TAL-T.
  Other Names: TAL-T; TAL-T cells
Drug: Serplulimab Injection — Srulizumab injection was given intravenous infusion both before and after the TAL-T cells infusion.

SUMMARY:
A Phase I clinical trial of the safety and tolerability of tumor-associated lymph node T cell injection in patients with advanced malignant solid tumors, including but not limited to melanoma, head and neck tumors, cervical cancer, and non-small cell lung cancer.

DETAILED DESCRIPTION:
The study was divided into two phases, the dose-range exploration study and the expanded enrollment study.

Exploration of the dosage range phase and the expanded enrollment phase were designed to evaluate the safety, tolerability, and initial efficacy of TAL-T cell therapy in patients with advanced solid tumors

ELIGIBILITY:
Inclusion Criteria:

1. Sign a written informed consent (ICF) and be able to comply with the visit and related procedures required by the program;
2. Age ≥18 years old, and ≤75 years old, male and female;
3. ECOG score 0-1;
4. Expected survival is not less than 12 weeks;
5. Advanced malignant solid tumors confirmed by cytology or histopathology (tumor markers combined with imaging can be used for some special advanced tumors, such as liver cancer) that have failed standard treatment or lack effective treatment methods, including but not limited to melanoma, head and neck tumors, cervical cancer, non-small cell lung cancer, etc.

   "Standard treatment failure" refers to the occurrence of disease progression after enough treatment courses and sufficient lines of treatment with the existing standard recommended therapy (refer to the latest CSCO guidelines), or recurrence after the regression of the tumor after standard treatment, or the toxic side effects of standard treatment are not tolerated.
6. There are tumor-associated lymph nodes that can be resected and T cells can be isolated: the tissue taken is ≥1 cm3, and the site has not received local treatment or has progressed after local treatment;
7. After sampling, subjects still have at least one evaluable lesion (Extended enrollment phase according to RECIST v1.1, subjects still have at least one measurable lesion (lesions that have received local treatment such as radiotherapy, interventional therapy, etc., cannot be considered as measurable lesions unless imaging evidence confirms clear progression of the lesion). That is, CT or MRI examination of non-lymph node lesions with the longest diameter ≥10 mm, and/or lymph node lesions with a short diameter ≥15 mm);
8. The subject has sufficient organ and bone marrow function (no blood transfusion or hematopoietic stimulating factors can be received within 14 days prior to screening)
9. Fertile men and women of reproductive age must agree to use effective contraception from the time they sign the ICF until one year after cell transfusion, and women of reproductive age must have a negative blood pregnancy test at the time of screening.

Exclusion Criteria:

1. meningeal metastases, and/or active brain metastases;
2. Have previously received allogeneic bone marrow transplantation, organ transplantation or are waiting for transplantation;
3. HBsAg positive hepatitis B; HCV-Ab positive hepatitis C; Positive for human immunodeficiency virus (HIV) antibodies; Syphilis antibody positive; Cytomegalovirus (CMV) IgM antibody positive; Human herpesvirus type 4 (EBV) IgM positive; Human T-lymphocytophilic virus (HTLV-Ⅰ/Ⅱ) antibody positive;
4. Received any fluorouracil chemotherapeutic drugs or small molecule targeted drugs within 14 days or 5 half-lives (whichever is shorter) prior to pretreatment; Received any antitumor biologic or non-fluorouracil chemotherapeutic drugs within 28 days or 5 half-lives (whichever is shorter) prior to pretreatment; Received radical radiotherapy or extensive radiotherapy within 28 days prior to pretreatment (except local non-target palliative radiotherapy for symptom relief within 14 days prior to pretreatment); Received Chinese medicine/Chinese herbal medicine with anti-tumor indications and local interventional therapy within 14 days prior to pretreatment;
5. Adverse events resulting from previous antitumor therapy have not returned to grade 1 or baseline levels (except for alopecia, grade 2 peripheral neurotoxicity, hypothyroidism controlled by alternative therapy and other toxicities that the investigators judged to be of no safety risk);
6. Persons who had been immunized with live attenuated vaccine within 28 days prior to pretreatment, or who required live attenuated vaccine immunization during the study period;
7. Had major surgery within 28 days prior to pretreatment, or required major surgery during the study period;
8. Long-term (≥3 days) treatment with systemic corticosteroids (dose ≥10 mg/ day of prednisone or equivalent hormone) or other immunosuppressive agents, except for inhalation or local use, is required 7 days before the tumor-associated lymph node excision sampling or during the study period;
9. Subjects with active systemic infections requiring intravenous antibiotic treatment within 7 days prior to screening;
10. Patients with active or past autoimmune diseases that are likely to recurs, such as systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vasculitis, psoriasis, etc. (subjects with hypothyroidism requiring only thyroid hormone replacement therapy, and subjects with type 1 diabetes requiring only insulin replacement therapy can be enrolled);
11. Previous or current cases of interstitial lung disease, coniosis, radiation pneumonia, severe impairment of lung function, etc.;
12. Hepatic encephalopathy, hepatorenal syndrome or Child-Pugh grade B or more severe cirrhosis, liver failure;
13. Third space effusion with poor clinical control before screening, such as pleural fluid and ascites that cannot be controlled by drainage or other methods;
14. Have a history of severe cardiovascular and cerebrovascular disease
15. Patients with pulmonary embolism or severe deep venous thrombosis of lower extremities during screening, requiring interventional therapy such as inferior vena cava filter placement, or using therapeutic dose of anticoagulants;
16. Any CTCAE 5.0 immune-related adverse reactions (irAE) grade ≥3 during any prior immunotherapy;
17. Those with immune checkpoints (such as PD-1) for treatment of other contraindications;
18. Subjects are participating in other interventional clinical studies;
19. Pregnant or lactating women;
20. The investigator believes that the subjects have other conditions that may affect their compliance or are not suitable to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-02-13 (Actual); Primary Completion 2026-12-19 (Estimated); Study Completion 2027-12-19 (Estimated)

PRIMARY OUTCOMES:
AEs and SAEs | All aes and saes are to be collected from the time the pre-screened informed consent is signed until 54 weeks after cell retransfusion, unless the subject withdraws from the study early for any reason
  Incidence, severity and drug correlation of AEs and SAEs

SECONDARY OUTCOMES:
ORR | Two years
  The proportion of subjects receiving a confirmed optimal response of PR or above which was evaluation according to RECIST or iRECIST principles.
DCR | Two years
  The proportion of subjects whose response was assessed as CR, PR, or stable disease (SD) to the total number of subjects for which response could be assessed
DOR | Two years
  The first assessment of efficacy was CR or PR up to PD or the time of death from any cause
PFS | Two years
  The time from the beginning of preconditioning until disease progression (PD) or death from any cause
OS | Two years
  The time from the subject's pre-treatment until death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Gaungdong, China

IPD SHARING:
Plan to Share IPD: No